CLINICAL TRIAL: NCT00310089
Title: A Pilot Study to Evaluate The Effects of Neoadjuvant AZD2171, a VEGF Receptor Tyrosine Kinase Inhibitor With Docetaxel, Doxorubicin, and Cyclophosphamide Chemotherapy in Previously Untreated Locally Advanced Breast Cancer
Brief Title: AZD2171 and Combination Chemotherapy in Treating Women With Locally Advanced Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000466185; NCI-06-C-0057; NCI-7088; NCT00273923 (obsolete NCT alias)
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2007-01

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Filgrastim; pegfilgrastim; cediranib; Cyclophosphamide; Docetaxel; Doxorubicin; Neoadjuvant Therapy

INTERVENTIONS:
Biological: filgrastim
Biological: pegfilgrastim
Drug: cediranib maleate
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Other: laboratory biomarker analysis
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: AZD2171 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as doxorubicin, cyclophosphamide, and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving AZD2171 together with combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed and may kill more tumor cells.

PURPOSE: This randomized clinical trial is studying how well giving AZD2171 together with combination chemotherapy works in treating women with locally advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall pathologic complete response rate in women with previously untreated, locally advanced breast cancer treated with neoadjuvant AZD2171, doxorubicin hydrochloride, cyclophosphamide, and docetaxel.

Secondary

* Compare changes in pretreatment levels of pKDR after 1 course of AZD2171 vs no medication.
* Determine the number of patients who respond to combination therapy beginning with the second course of therapy.
* Determine the clinical response rate in patients treated with this regimen.
* Determine the safety of this regimen in these patients.
* Determine the changes in tumor proliferation (Ki67) in these patients.
* Determine the pharmacokinetics and pharmacogenetics of this regimen in these patients.
* Correlate angiogenic parameters with tumor response in these patients.
* Determine tumor vascularity and permeability before and after treatment as seen on dynamic contrast-enhanced MRI and initial area under the gadolinium curve.
* Determine tumor choline levels before and after treatment as measured by quantitative single-voxel MR spectroscopy and correlate with response.

OUTLINE: This is a multicenter, randomized, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral AZD2171 once daily on days 1-7* during course 1. During the second and subsequent courses, patients receive oral AZD2171 once daily on days 1-21, doxorubicin hydrochloride IV over 3-5 minutes, cyclophosphamide IV over 30 minutes, and docetaxel IV over 1 hour on day 1. Patients also receive filgrastim (G-CSF) subcutaneously (SC) on days 2-11 or pegfilgrastim SC on day 2. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *If biopsy cannot be scheduled prior to day 7 or 8 of course 1, AZD2171 alone can be continued for up to 14 days.

* Arm II (control): Beginning during the second course, patients receive AZD2171, doxorubicin hydrochloride, cyclophosphamide, docetaxel, and G-CSF or pegfilgrastim as in arm I.

All patients undergo tumor biopsiesat at baseline, before courses 2 and 4, and 3 weels after completion of study treatment. Tissue is examined for various biomarkers (phosphorylated-KDR, -MAPK, and -Akt, Ki67, VEGF, and p53) and for DNA ploidy analysis**.

NOTE: **Patients also undergo dynamic contrast-enhanced MRI and quantitative magnetic resonance spectroscopy 1 week before beginning therapy, 24 hours after starting therapy, prior to courses 2, 4, and 6, and 3 weeks after completion of study treatment.

After completion of AZD2171 and chemotherapy, patients undergo surgical resection.

After completion of study treatment, patients are followed for 4 weeks.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer, meeting 1 of the following criteria:

  * Previously untreated disease
  * Inflammatory disease
  * Locally advanced breast cancer (stage IIIA, IIIB, or IIIC disease)
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion (longest diameter) ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan or breast MRI
* Accessible tumor tissue for serial biopsy
* No overexpression of HER2
* No known brain metastases secondary to breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Karnofsky performance status 60-100%
* Life expectancy > 3 months
* Female only
* Menopausal status not specified
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8 g/dL
* Bilirubin normal (≤ 2 times upper limit of normal [ULN] if evidence of Gilbert's disease and elevated bilirubin not related to tumor or other liver disease)
* AST and ALT ≤ 2.5 ULN
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Proteinurea ≤ +1 on 2 consecutive dipsticks at least 1 week apart
* INR ≤ 1.5
* LVEF ≥ 50% by MUGA or echocardiogram without clinical symptoms or signs of heart failure
* Fertile patients must use effective contraception
* Not pregnant or nursing
* Negative pregnancy test
* No peripheral neuropathy ≥ grade 2
* No known CNS disease, including history of stroke or seizures not controlled by standard medical therapy
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel, doxorubicin hydrochloride, or cyclophosphamide
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Hypertension
  * Ongoing or active infection requiring IV antibiotics
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Peripheral vascular disease ≥ grade II
  * Psychiatric illness/social situation that would preclude study treatment
* No nonhealing wounds or bone fractures within the past 28 days
* No history of an active malignancy except carcinoma in situ of the cervix or nonmelanomatous skin cancer in the past 5 years

PRIOR CONCURRENT THERAPY:

* No prior surgery, chemotherapy, or hormonal therapy for breast cancer
* No concurrent medication that may affect renal function (e.g., amphotericin B or pentamidine)
* No full-dose oral or parenteral anticoagulants or chronic daily treatment with aspirin (dose > 325 mg/day) within the past 10 days
* No other concurrent investigational agents
* No other concurrent commercially available drugs for this cancer
* No concurrent antiretroviral therapy for known HIV infection
* No major surgery within the past 28 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2006-01; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neelima Denduluri, MD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey